CLINICAL TRIAL: NCT05958706
Title: Mitochondrial Substrate Utilization in the Diabetic Human Heart
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-1962
Record Dates: First submitted 2023-07-03; First posted 2023-07-25 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Heart Failure; Type2diabetes; Insulin Resistance; Mitochondrial Diseases; Diabetic Cardiomyopathies
Keywords: mitochondrial function; respirometry; heart failure; type 2 diabetes mellitus; insulin resistance; mitochondrial disease; diabetic cardiomyopathy
MeSH Terms: conditions — Heart Failure; Insulin Resistance; Mitochondrial Diseases; Diabetic Cardiomyopathies; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- patients with manifest heart failure: patients with manifest heart failure and T2DM or patients with manifest heart failure without T2DM
- patients with terminal heart failure: patients with terminal heart failure and T2DM or patients with terminal heart failure without T2DM
- patients after heart transplantation: patients after heart transplantation and T2DM or patients after heart transplantation without T2DM

SUMMARY:
Diabetes can lead to heart failure independently, but the underlying causes remain incompletely understood. The main aim of this study is to identify differential regulation of mitochondrial substrate utilization and complex activity in heart failure and type 2 diabetes mellitus (T2DM). For this, we will conduct a prospective, observational study to examine myocardial mitochondrial oxidative function and related metabolic parameters, gene expression, histological markers, and inflammation in cardiac tissue from patients with heart failure or patients after heart transplantation. We will further assess cardiac function using cardiac magnetic resonance imaging with and without stress protocols and magnetic resonance spectroscopy. Glycemic control/T2DM will be characterized by oral glucose tolerance tests. The results of this project will help to better understand the cellular mechanisms of the development of diabetic cardiomyopathy and contribute to the development of early diagnostic, as well as therapeutic approaches for the prevention and treatment of diabetic cardiomyopathy.

DETAILED DESCRIPTION:
Insulin resistance, ectopic lipid accumulation in the liver, and plasma concentrations of free fatty acids are independent predictors of cardiac mortality, the primary cause of death in patients with type 2 diabetes mellitus (T2DM). T2DM predisposes to the development of heart failure independently of other risk factors. Ventricular dysfunction in diabetic patients independent of coronary artery disease or arterial hypertension is termed diabetic cardiomyopathy. Studies suggest that myocardial mitochondrial dysfunction, as well as accumulation of lipids and other metabolites, oxidative stress, and altered insulin signaling, play a significant role in the pathogenesis of diabetic cardiomyopathy. Thus, we also found evidence of impaired mitochondrial function in hyperglycemia and insulin resistance in previous analyses. Nevertheless, it remains unclear, among other things, at which point of mitochondrial metabolism the shown impairments originate, whether the availability of different substrates may influence these effects, what is the temporal sequence of pathomechanistic events, and what are the effect modifiers for the influence of T2DM on the myocardium.

The goal of the present work is to more precisely characterize the underlying pathomechanisms to answer these questions. The focus will be on respirometric analysis of human myocardial tissue samples established by our preliminary work. In previously published studies, we were able to establish its use for the first time in catheter-guided endomyocardial biopsies. By studying further heart failure and heart transplant patients, we will analyze the importance of myocardial mitochondrial function as a prognostic marker of further disease progression and, using larger power, investigate the influence of different effect modifiers.

The results of this project will help to better understand the cellular mechanisms of the development of diabetic cardiomyopathy and contribute to the development of early diagnostic, as well as therapeutic approaches for the prevention and treatment of diabetic cardiomyopathy.

Hypotheses:

1. the reduced mitochondrial oxidative capacity of myocardial mitochondria in T2DM is complex- and substrate-specific.
2. within patients with heart failure of unclear etiology and indication for myocardial biopsy, there are mitochondrial profiles with different clinical courses and outcomes.
3. in T2DM, myocardial oxidative capacity is also longitudinally impaired in heart transplant patients and this impairment is associated with worse clinical outcome.

Objectives:

1. identify specific targets for therapeutic strategies against diabetic cardiomyopathy: work program (WP) 1.
2. characterization of myocardial mitochondrial function and its relevance to clinical phenotypes in heart failure: WP 2.
3. investigation of T2DM as a longitudinal predictor of worse mitochondrial and clinical cardiac function in heart transplant patients: WP 3.

WP1:

The aim is to identify altered respiratory chain subcomponents and metabolic pathways associated with the development of manifest diabetic cardiomyopathy in T2DM. For this purpose, patients with and without T2DM (according to the criteria of the "American Diabetes Association" (ADA)) who have an indication for endomyocardial biopsy on clinical grounds will be included. A matched comparison between patients with and without T2DM will provide evidence of diagnostic and therapeutic targets for diabetic cardiomyopathy in newly diagnosed heart failure (with and without left ventricular ejection fraction limitation).

Patients:

* Group 1: Patients with manifest heart failure (NYHA II-IV) with clinical indication to perform myocardial biopsy and T2DM according to the "American Diabetes Association" (ADA) criteria, HbA1c < 9.0%, with/without therapy (insulin, oral/parenteral antidiabetic drugs).
* Group 2: Patients with manifest heart failure (NYHA II-IV) with clinical indication to perform myocardial biopsy without T2DM.

WP2:

The aim is to characterize myocardial mitochondrial function and its relevance for clinical phenotypes in heart failure. For this purpose, patients with terminal heart failure from the heart failure program of the Department of Cardiology, Pneumology and Angiology of the University Hospital Düsseldorf who are scheduled for implantation of a left ventricular assist device (LVAD) or are undergoing heart transplantation will be included.

All study examinations of myocardial tissue are performed in an area of the left ventricular apex obtained during surgery (LVAD implantation or cardiac harvest), which is not further clinically analyzed or preserved and which therefore no longer has any direct benefit for the patients.

Patients:

* Group 1: Patients with terminal heart failure and diagnosed T2DM according to the "American Diabetes Association" (ADA) criteria 18, HbA1c < 9.0%, with/without therapy (insulin, oral/parenteral antidiabetic drugs).
* Group 2: Patients with terminal heart failure (NYHA IV) without T2DM.

WP3:

The aim is to investigate T2DM as a longitudinal predictor of impaired mitochondrial and clinical cardiac function in heart transplant patients. For this purpose, patients who are included in the heart transplantation follow-up program of the University Hospital Düsseldorf and have the indication for endomyocardial biopsy within this program will be included. Routine myocardial biopsy is necessary in these patients to detect subclinical graft rejection early, as it is associated with increased mortality. Biopsies occur multiple times in the first year after transplantation, and in subsequent years (if there is no evidence of rejection), the goal is to monitor annually.

Patients:

* Group 1: Patients after heart transplantation with diagnosed T2DM according to the "American Diabetes Association" (ADA) criteria 18, HbA1c < 9.0%, with/without therapy (insulin, oral/parenteral antidiabetic drugs).
* Group 2: Patients after heart transplantation without T2DM.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 20 and ≤ 85 years
* Male and female patients with manifest heart failure (NYHA II-IV) and clinical indication for myocardial biopsy or after transplantation and clinical indication for myocardial biopsy with or without type II diabetes mellitus or terminal (NYHA IV) heart failure with or without type II diabetes mellitus.
* Written informed consent

Exclusion Criteria:

* Acute infectious diseases within the last 2 weeks before the examination
* Autoimmune diseases or acute immunocompromising diseases (leukocytes < 5000/μl)
* Pregnancy
* Use of alcohol or drugs (addiction), psychiatric diseases
* Suspected or manifest AIDS (HIV); hepatitis B or C.
* Liver disease not attributed to the presence of nonalcoholic fatty liver hepatitis or congestive hepatopathy in heart failure
* Malignant cancer
* Lack of capacity to give informed consent or lack of consent to participate in the study
* For MRI study with drug stress: contraindications to the use of regadenoson, specifically: a) Hypersensitivity to the active ingredient or any of the other ingredients mentioned. b) Second- or third-degree atrioventricular (AV) block or sinus node dysfunction, unless these patients have a functioning pacemaker. c) Unstable angina that has not been stabilized with medication. d) Severe hypotension. e) Decompensated stages of heart failure.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with heart failure with or without T2DM undergoing endomyocardial biopsy for clinical reasons (WP1), patients with terminal heart failure with or without T2DM undergoing left ventricular assist device surgery or heart transplantation (WP2), and patients after heart transplantation with and without T2DM undergoing endomyocardial biopsy for clinical reasons (post-transplant surveillance).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Substrate-specific JVO2 of ventricular myocardial mitochondrial oxidative capacity | at time of the endomyocardial biopsy procedure
  measured in (pmol/s*mg)

SECONDARY OUTCOMES:
Markers of cardiac function and structure | 1 day before or after endomyocardial biopsy
  measured by cardiac magnet resonance tomography
Markers of cardiac function | 1 day before or after endomyocardial biopsy
  measured by echocardiography
Cardiac substrate utilization | 1 day before or after endomyocardial biopsy
  measured by cardiac magnet resonance spectroscopy (MRS)
Patterns in the myocardial transcriptome and systemic metabolome | at time of the endomyocardial biopsy procedure
non-fatal myocardial infarction | up to 5 years (follow-up in clinical routine)
  Survival and clinical outcomes after study index visit (inclusion)
all-cause mortality | up to 5 years (follow-up in clinical routine)
  Survival and clinical outcomes after study index visit (inclusion)
allograft rejection | up to 5 years (follow-up in clinical routine)
  Survival and clinical outcomes after study index visit (inclusion)
hospitalization for heart failure | up to 5 years (follow-up in clinical routine)
  Survival and clinical outcomes after study index visit (inclusion)
non-fatal stroke | up to 5 years (follow-up in clinical routine)
  Survival and clinical outcomes after study index visit (inclusion)
Longitudinal Substrate-specific JVO2 | variable, up to 2 years
  measured with sequential biopsies

CONTACTS AND LOCATIONS:
Overall Officials: Malte Kelm, Prof., Study Chair — Clinic for Cardiology, Pneumology and Angiology at University Hospital Düsseldorf; Daniel Scheiber, MD, Principal Investigator — Clinic for Cardiology, Pneumology and Angiology at University Hospital Düsseldorf
Locations (1):
- University-Hospital Düsseldorf Division of Cardiology, Pulmonary Disease and Vascular Medicine, Düsseldorf, Germany

IPD SHARING:
Plan to Share IPD: No